CLINICAL TRIAL: NCT06906913
Title: Evaluation of Oropharyngeal and Anal Swab Samples in Patients With HPV Positivity
Brief Title: Oral and Anal Swab Sampling in Patients With HPV Positivity
Acronym: Oral Anal HPV
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Collaborators: gaziantep university medicine faculty (Unknown)
Responsible Party: Principal Investigator, Tugba Akcaoglu, Doctor of Medicine, Medipol University
Other Study IDs: Number 362; TF.HZP.23.31 (Other Grant/Funding Number: Gaziantep University Scientific Research Project support program)
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: HPV
Keywords: Anal; cervical; human papillomavirus; oropharyngeal; screening

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — Oropharyngeal and anal swab samples will be obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Swab Sampling: Oropharyngeal and anal swab samples are obtained.
  Interventions: Diagnostic Test: HPV testing

INTERVENTIONS:
Diagnostic Test: HPV testing — Oropharyngeal and anal swab samples are evaluated in the Microbiology laboratory for the existence of HPV.

SUMMARY:
Patients whose pathology results are reported as cervical intraepithelial neoplasia (CIN) 1, CIN 2, and CIN 3, are recruited. We aimed to evaluate HPV-positive women presenting to the Obstetrics and Gynecology clinic, whose cervical pathology results were reported as CIN 1, CIN 2, and CIN 3, by collecting oropharyngeal and anal swab samples. A total of 30 women of reproductive age, who consented to participate, were included in the study.

DETAILED DESCRIPTION:
Human papillomavirus (HPV) positivity is associated with cervical, oropharyngeal, and anal cancers. There is insufficient data in the current literature regarding the effectiveness of obtaining oropharyngeal and anal swabs from patients with HPV positivity is an effective method for detecting potential pathologies. HPV-positive women presenting to the Obstetrics and Gynecology clinic, whose cervical pathology results were reported as CIN 1, CIN 2, and CIN 3, will be evaluated by collecting oropharyngeal and anal swab samples.

ELIGIBILITY:
Inclusion Criteria:

* HPV-positive women presenting to the Obstetrics and Gynecology clinic, whose cervical pathology results were reported as CIN 1, CIN 2, and CIN 3

Exclusion Criteria:

* HPV-negative women

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Study Population: A total of 30 women of reproductive age, who consented to participate, will be included in the study.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal Swab Sample - HPV Testing | 1 month
  Presence of HPV will be tested
Anal Swab Sample - HPV Testing | 1 month
  Presence of HPV

SECONDARY OUTCOMES:
Oropharyngeal Swab Sample - HPV Testing (if positive) | 1 month
  Type of HPV
Anal Swab Sample - HPV Testing (if positive) | 1 month
  Type of HPV

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Bayramoglu Tepe, Doctor of Medicine, Study Director — University of Gaziantep; Ozan Dogan, Prof. Dr., Study Chair — Istanbul Nisantasi University
Locations (1):
- Gaziantep Cengiz Gokcek Women's, Obstetrics and Pediatrics Hospital, Gaziantep, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The study results can be kept confidential before being published in a journal.